CLINICAL TRIAL: NCT03910413
Title: Dual Energy CT as a Noninvasive Method to Screen for Gastroesophageal Varices
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended and enrollment challenged by COVID and other factors.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Andrew Dennis Smith, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R18-098
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Gastroesophageal Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dual Energy CT (Other)
  Interventions: Diagnostic Test: Duel Energy CT

INTERVENTIONS:
Diagnostic Test: Duel Energy CT — Enrolled subjects will complete a dual energy ct for evaluation of esophageal varices

SUMMARY:
Cirrhosis leads to portal hypertension and development of gastroesophageal varices, which are the most common cause for bleeding in cirrhosis and a major cause of death. The American Association for the Study of Liver Disease (AASLD) recommends screening endoscopy every 2 years to evaluate for gastroesophageal varices, and annual surveillance for those with small varices on endoscopy. Unfortunately, endoscopy is costly, requires sedation, is poorly tolerated, is subject to high inter-observer variability, and is associated with risks that include bleeding, esophageal injury and aspiration. Noninvasive methods for evaluation of gastroesophageal varices are needed. CT is noninvasive, rapid, less expensive than endoscopy, requires no sedation, provides a quantitative measure of the size of the varices, and allows for assessment of para-esophageal varices, varices in other body locations, ascites, other signs of portal hypertension, patency of liver vasculature, and detection, diagnosis and staging of hepatocellular carcinoma. Single-Energy CT (SECT) has relatively high accuracy in prospective studies for detection of any and large varices but is associated with suboptimal contrast opacification of gastroesophageal varices. Dual-Energy CT with the GE scanners with GSI Xtream (DECT) improves the contrast-to-noise ratio by 60% compared to SECT and is currently standard of care at UAB for evaluation of cirrhosis. The primary objective of this study is to determine the accuracy of DECT for detecting any varices and high-risk varices. The study hypothesis is that the accuracy (AUROC) of DECT will be >0.90 and >0.95 for detecting any and high-risk varices in a prospective pilot study (N=50) that uses endoscopy as the reference standard. This will be a single-center pilot observational prospective IRB-approved study. A total of 50 adult patients presenting to UAB Endoscopy for surveillance endoscopy to detect and grade gastroesophageal varices will be enrolled.

DETAILED DESCRIPTION:
Cirrhosis leads to portal hypertension and development of gastroesophageal varices, which are the most common cause for bleeding in cirrhosis and a major cause of death. Bleeding varices have a 6-week mortality of 15%-25%. About 50% of patients with cirrhosis have varices, and 30% have large varices (>5 mm) that are high risk for bleeding.

The American Association for the Study of Liver Disease (AASLD) recommends screening endoscopy every 2 years to evaluate for varices, and annual surveillance for those with small varices on endoscopy. Patients at a high risk of bleeding with large varices, small varices and red wale signs (an endoscopic finding), or small varices and decompensated cirrhosis proceed to treatment such as prophylactic band ligation and beta blockers. Conversely, patients with no varices or small varices (≤5 mm) continue surveillance efforts by endoscopy to monitor for development of large varices. Unfortunately, endoscopy is costly, requires sedation, is poorly tolerated, is subject to high inter-observer variability, cannot detect other signs or portal hypertension or para-esophageal varices that are at risk for future bleeding events, and is associated with risks that include bleeding, esophageal injury and aspiration. Many of these factors contribute to poor patient compliance with AASLD recommendations.

Noninvasive methods for detecting, grading, and risk stratification of esophageal varices are needed. Imaging tests such as ultrasound elastography to measure liver stiffness have been proposed as a method to predict the presence of varices but have insufficient accuracy to eliminate the need for endoscopy.10 An ideal biomarker to screen for esophageal varices would be part of the routine standard of care of patients with cirrhosis, noninvasive, rapid, less expense than endoscopy, highly accurate, highly reproducible, and would require no sedation, provide a quantitative measure of the size of the varices, provide a mechanisms to assess the risk of future bleeding, allow for an assessment for other signs of portal hypertension, and provide other benefits to the patient (e.g. detect ascites and HCC and assess liver vasculature).

Computed tomography (CT) is standard of care to screen for HCC. CT is noninvasive, rapid, less expensive than endoscopy, requires no sedation, provides a quantitative measure of the size of the varices, and allows for assessment of para-esophageal varices, varices in other body locations, ascites, other signs of portal hypertension, patency of liver vasculature, and detection, diagnosis and staging of HCC. Conventional Single-Energy CT (SECT) has relatively high accuracy in prospective studies for detection of any and large varices and has higher inter-observer agreement than endoscopy (kappa 0.56 vs. 0.36, respectively). Major deficiencies in SECT include relatively suboptimal contrast opacification of gastroesophageal varices, inconsistent accuracy that is dependent upon SECT image acquisition technique, and suboptimal stratification of the risk of bleeding (e.g. inability to detect red wale sign) compared to endoscopy.

Dual-Energy CT (DECT) improves the contrast-to-noise ratio by 60% compared to SECT. DECT also improves visualization by taking advantage of the markedly increased attenuation of iodine at photon energy levels just above the iodine K edge (33 keV). Using material decomposition techniques, DECT can map the concentration of iodine on a voxel by voxel basis which, combined with higher contrast to noise resolution on these same type of images, improves the conspicuity of enhancing structures. DECT is routinely used to screen for HCC in cirrhotic patients.

While DECT has been shown to improve image quality and portal venography compared to SECT, the accuracy of DECT for screening for varices has not been reported. The primary objective is to determine the accuracy of dual energy CT for detecting any varices and high-risk varices in patients with cirrhosis presenting for upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with cirrhosis presenting to UAB Endoscopy for surveillance endoscopy to detect and grade gastroesophageal varices

Exclusion Criteria:

* Inability to provide written informed consent
* History of bleeding gastroesophageal varices, variceal intervention or portosystemic shunt
* Prior liver transplant
* History of malignancy
* Severe chronic kidney disease with estimated glomerular filtration rate (GFR) < 30 mL/min/1.73 m2
* Presence of acute kidney injury
* Prior iodinated contrast allergy
* Patient weight >300 lbs
* Multiphasic liver CT within 3 months of upper endoscopy
* Pregnancy
* Inclusion of all races and ethnic groups are eligible for this trial. There is no bias towards age or race in this trial. The trial is open the accrual of women and men.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital Outpatient Imaging, Leeds and Gardendale locations, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dual Energy CT
Started | 11
Completed | 6
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dual Energy CT
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 59 [31 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Measure the Accuracy of Dual Energy CT for Detecting Any Varices and High-risk Varices in Patients With Cirrhosis Presenting for Upper Gastrointestinal Endoscopy.
Description: Varices on dual energy CT will be graded as follows: 0 = no varices, 1 = small [<5 mm] varices, and 2 = large / high risk [>= 5 mm] varices. The reference standard for this outcome will be grading of varices on endoscopy (0 = no varices, 1 = small (< 5 mm) varices, and 2 = large (>=5 mm) varices.
Time Frame: DECT will be no more than 2 weeks from the time of endoscopy
Population: The study was ended prematurely due to covid. This data was not collected.
Arm/Group | Dual Energy CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Dual Energy CT
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03910413/Prot_SAP_000.pdf